CLINICAL TRIAL: NCT07344155
Title: SOAR: Surgery Objective Analysis and Review
Acronym: SOAR
Status: Not yet recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Wellcome Trust (Other); Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00487162
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Surgical Education and Skill Acquisition
Keywords: surgical education

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SOAR Webapp: surgical residents through all years of training
  Interventions: Other: SOAR Webapp-Based Video Review and Feedback

INTERVENTIONS:
Other: SOAR Webapp-Based Video Review and Feedback — Surgical residents will use the SOAR Webapp, a video-based surgical education platform, to review intracorporeal laparoscopic procedure recordings and receive structured feedback on technical skills and surgical decision-making. The intervention includes post-operative video review with an expert surgeon and automated analytic outputs generated by computer vision algorithms, including performance metrics and annotated video segments. The intervention is used for educational and training purposes only and does not alter patient care.

SUMMARY:
The purpose of this pilot study is to determine the feasibility and usability of a surgical software training platform called the SOAR Webapp that will allow Johns Hopkins surgical trainees to receive rapid qualitative and quantitative feedback on both technical skills and surgical decision-making. The SOAR Webapp is a software device comprised of artificial intelligence (AI) computer vision algorithms embedded in a standalone mobile application. The software will be able to take laparoscopic videos as input and output the automated assessments for users. The investigators will also set up the clinical and logistical infrastructure needed to conduct a pilot study to evaluate the effectiveness of the SOAR computer vision system in facilitating video-based review of trainee performed operations with feedback from an expert attending surgeon. The investigators hypothesize that the video review features of the SOAR Webapp will be an effective training aid and has the potential to improve surgical education and training.

ELIGIBILITY:
Inclusion Criteria:

Surgery Residents:

* General surgery trainee or attending surgeon at Johns Hopkins.
* Must be able to operate.
* 18 years or older

Patients:

* Undergoing laparoscopic surgery at Johns Hopkins

Exclusion Criteria:

* None for surgery residents
* Patients: cases without record of video

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be general surgery residents at Johns Hopkins University School of Medicine. All residents from all post graduate training years will be able to participate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Perceived resident educational impact and accuracy of operative performance assessment as measured by the SOAR Post-Intervention Evaluation Survey | 2 years
  This is a survey completed by surgical trainees following use of the SOAR Web Application. The survey evaluates trainee perceptions of:
  * Engagement in deliberate practice behaviors
  * Accuracy and usefulness of operative performance assessments (including psychomotor skill, tissue handling, operative progress, exposure quality, dissection quality, and error detection)
  * Accuracy and usefulness of pre-populated operative steps
  * Impact of the SOAR Web Application on the frequency and quality of engagement with attending surgeons
  * Overall usability and perceived challenge of the SOAR Web Application
  All survey items are measured using a 3-point Likert scale (Never, Sometimes, Often), with higher scores indicating greater perceived frequency, accuracy, usefulness, or educational impact, depending on the item. Survey responses are analyzed at the individual item level and summarized as frequencies and proportions. The maximum score is 30, minimum 10.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey K Jopling, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No